CLINICAL TRIAL: NCT00715013
Title: Patupilone (EPO 906) in Patients With Recurrent or Progressive Glioblastoma Multiforme Prior to and After Secondary Resection: an Open-label Phase I/II Trial.
Brief Title: Patupilone (EPO 906) in Patients With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2401
Record Dates: First submitted 2007-11-22; First posted 2008-07-14 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-08

CONDITIONS: Recurrent Glioblastoma Planned for Reoperation
Keywords: recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — epothilone B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Patupilone — Patupilone

SUMMARY:
Patupilone trial for patients with recurrent glioblastoma, which are planned for re-operation. Objectives: prolongation of PFS compared to patients with re-operation only, Patupilone tumor concentrations, pharmacokinetic, Perfusion in MRI pre - and post Patupilone. Translational research of tumor tissue exposed to patupilone.

* Trial with medicinal product

DETAILED DESCRIPTION:
Prior to and after re-operation patients with recurrent glioblastoma receive the investigational drug Patupilone, a tubulin-inhibitor.

The purpose of the trial is to prolong PFS in this patient population. Patupilone is already used in clinical trials of other tumor entities such as ovarian cancer, breast and lung cancer. Side effects are expected to be manageable.

ELIGIBILITY:
Inclusion criteria:

* Recurrent glioblastoma at least 2 cm in diameter after standard treatment (Surgery, Radiotherapy and Chemotherapy), which has to be completed at least three weeks earlier.
* > 18 years of age, KPS 70-100%
* No liver disease, no malignancies (except curative treated skin tumors, DCIS of the breast and curative treated cervix carcinoma)
* Lc > 3000 und Tc > 100 000, Hb> 9, Bilirubin </= 1.5mg/dl, AST/ALT less than 2.5 x upper limit, creatinine </= 132umol/l
* No pregnancy or breast feeding
* Written Informed Consent prior to study entry
* No reasons for incompliance
* Reoperation planned

Exclusion criteria:

* KPS < 70%
* Radiotherapy- or Chemotherapy within 6 weeks
* Enzyme inducing medication or St John's wort
* Other study medication within 28 days
* Other malignancies
* Intolerance of Patupilone
* Prior Patupilone
* Neuropathy > Grad 1
* Other life threatening illnesses
* Acute or chronic liver diseases
* HIV Infection
* Known non-compliance in medication intake,inability to give informed consent
* Cardiac problems (NYHA III oder IV) with uncontrolled insufficiency or angina pectoris
* Active or uncontrolled infection
* Pregnancy or breast feeding
* Hematologic Growth Factors (without Erythropoetin) colostomy
* Patients with uncontrolled diarrhea in the last 7 days prior to study entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years
PFS, OS translational research | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Hofer, MD, Principal Investigator — UniversitaetsSpital Zuerich